CLINICAL TRIAL: NCT01403909
Title: Effect of Pneumatic Intermittent Venous Compression on Fluid Volumes Infused During Major Abdominal Surgery in Non-obese American Soceity of Anesthesiologists (ASA) 1-3 Patients
Brief Title: Effect of Pneumatic Intermittent Venous Compression on Fluid Volumes Infused During Major Abdominal Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We need somebody to replace the principal inestigator.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LOCAL/2011/DC-04; 2011-A00800-41 (Other: RCB number)
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Major Abdominal Surgery
MeSH Terms: interventions — Intermittent Pneumatic Compression Devices; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With compression (Experimental): The patients randomized to this group will have intermittent pneumatic venous compression of the lower limbs during surgery.
  Interventions: Device: Intermittent pneumatic compression
- Without compression (Active Comparator): The patients randomized to this group will not have intermittent pneumatic venous compression of the lower limbs during surgery. (Standard care)
  Interventions: Procedure: Standard care

INTERVENTIONS:
Device: Intermittent pneumatic compression — Intermittent pneumatic venous compression is applied to the lower limbs of patients during surgery.
  Arms: With compression
Procedure: Standard care — Intermittent pneumatic venous compression is not applied to the lower limbs of patients during surgery.
  Arms: Without compression

SUMMARY:
The main objective of this study was to evaluate the effect of intermittent pneumatic venous compression on intra-operative fluid intake by comparing two groups of patients with or without intermittent pneumatic compression of the lower limbs.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Patient with ASA score 1-3
* Body mass index < 30 kg/m^2
* Patient is schelduled for major abdominal surgery (laparotomy without risk of haemorrhage whose duration is assumed to be greater than 120 min)
* The patient passes from home, directly to the hospital, without schelduled hospitalization in another department

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant
* The patient is breastfeeding
* The patient has a contra-indication for treatment necessary for the study
* ASA score > 3
* body mass index > 30 kg/m^2
* Expected surgical time of < 120 minutes
* Surgery with risk of hemorrhage
* Surgery via celioscopy
* The surgery require perineal access, thus rendering any blinding impossible
* Hepatic surgery
* Contra indication for intermittent venous compression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Volume fluids (ml) | End of surgery (expected mean of 2 hours)
  The total volume of infused fluids (Ringer's Lactate and HES) delivered to the patient during surgery (ml)

SECONDARY OUTCOMES:
Hypotensive episodes | end of surgery (expected mean of 2 hours)
  The number of arterial hypotension episodes (systolic pressure < 90 mmHg)
VEGF | end of surgery (expected mean of 2 hours)
  Concentration (pg/ml) of Vascular Endothelial Growth Factor (VEGF) in blood
sFlt1 | end of surgery (expected mean of 2 hours)
  Concentration (pg/ml) of soluble vascular endothelial growth factor receptor-1 (sFlt1) in blood
Hematocrit % | end of surgery (expected mean of 2 hours)
Albumin | end of surgery (expected mean of 2 hours)
  Albuminemia (g/l)
Prothrombin (%) | end of surgery (expected mean of 2 hours)
  Prothrombin rate in blood
Activated partial thromboplastin time | end of surgery (expected mean of 2 hours)
  Activated partial thromboplastin time (seconds)
Presence/absence of POSSUM complications | 28 days
  Presence/absence of complications as defined by the Physiological and Operative Severity Score for the Enumeration of Mortality and Morbidity (POSSUM) criteria
Days of hospitalization | 28 days
  Length of hospitalization (days)
Number of days not in hospital | 28 days
  Number of days not in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Damien Candela, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France